CLINICAL TRIAL: NCT00393757
Title: Malaria Transmission and Immunity in Highland Kenya
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0124; NCT00776061 (obsolete NCT alias)
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2007-10

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Malaria, Plasmodium falciparum, Kenya
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to see why malaria epidemics occur in highland areas in Kenya. A better understanding of factors contributing to malaria may be necessary for malaria vaccine planning. These factors include interactions between age, where malaria is passed from mosquitoes to people, immune system (how the body fights infection) responses and other factors that contribute to malaria in epidemic-prone areas. About 6400 people from the villages of Kapsisiywa and Kipsamoite will participate. Study procedures will include in home surveys, which will involve a census and an interview by researchers. Blood samples and smears will be collected from some volunteers in both communities to understand how the body protects itself from malaria and to check for malaria parasites. Twice each month, random houses will be selected from 3 places in the village to measure the number of mosquitoes in the home. Participants may be involved in the study for up to 4 years.

DETAILED DESCRIPTION:
The purpose of this study is to see why malaria epidemics occur in highland areas in Kenya. A better understanding of factors contributing to malaria may be necessary for malaria vaccine planning. These factors include interactions between age, where malaria is passed from mosquitoes to people, immune system (how the body fights infection) responses and other factors that contribute to malaria in epidemic-prone areas. About 6400 people from the villages of Kapsisiywa and Kipsamoite will participate. Study procedures will include in home surveys, which will involve a census and an interview by researchers. Blood samples and smears will be collected from some volunteers in both communities to understand how the body protects itself from malaria and to check for malaria parasites. Twice each month, random houses will be selected from 3 places in the village to measure the number of mosquitoes in the home. Participants may be involved in the study for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

Active surveillance of clinical malaria -Individuals of any age who live in the area (Kipsamoite or Kapsisiywa) for more than 6 months of the year, or, if they are new to the area, who plan to live in the area for more than 6 months of the year (permanent residents).

Passive surveillance of clinical malaria

-Any individual living within the boundaries of the 2 study areas (Kipsamoite and Kapsisiywa)

Exclusion Criteria:

Active surveillance of clinical malaria

* Declining to participate in the study
* Will be gone from site more than 1 week per month
* Not available for weekly symptom check or bimonthly blood sample collection

Passive surveillance of clinical malaria

* Declining to participate in the study
* Participation in active surveillance study

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20610
Dates: Start 2006-10; Primary Completion 2011-01-31 (Actual); Study Completion 2011-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya